CLINICAL TRIAL: NCT06495229
Title: A Multicenter, Single Arm, Open Label Study to Evaluate the Safety and Efficacy of CM310 in Adolescent Patients With Atopic Dermatitis
Brief Title: Study of CM310 in Adolescent Subjects With Atopic Dermatis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310-101215
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 group (Experimental)
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — Interleukin-4 receptor(IL-4Rα) monoclonal antibody

SUMMARY:
This is a multi-center, single arm, open label phase 3 study to evaluate the safety and efficacy of CM310 in children patients with moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the study and voluntarily sign a written informed consent form (ICF).
* Subjects who must complete the evaluation of Week 18 of the main study.
* With Atopic Dermatitis.

Exclusion Criteria:

* Any major surgery planned during the research period.
* Subjects with potential fertility do not agree to adopt efficient contraceptive measures throughout the entire study period; Pregnant or breastfeeding women, or women planning to conceive or breastfeed during the study period.
* With any circumstance that the subject is not suitable to participate in this study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to week 52
  Incidence of adverse events.

SECONDARY OUTCOMES:
Change from baseline in Eczema Area and Severity Index (EASI) | up to week 62
  Changes from baseline in Eczema Area and Severity Index (EASI)
Proportion of subjects with Immunoglobulin A(IGA) 0 or 1 and a reduction of from baseline of ≥ 2 points | up to week 62
  Proportion of subjects with IGA 0 or 1 (on a 5-point scale, range from 0-4 point, higher scores mean a worse disease severity) and reduction ≥2 points from baseline.
Improvement of Numerical Rating Scale (NRS) | up to week 62
  Proportion of subjects with improvement (reduction) of pruritus NRS from baseline. The range of NRS is from 0 (no itch)-10 (worst imaginable itch).
Body surface area (BSA) of involvement of atopic dermatitis | up to week 62
  Change from baseline in percent of BSA
Children Dermatology Life Quality Index (CDLQI) | up to week 62
  Changes from baseline in CDLQI
Patient-Oriented Eczema Measure (POEM) | up to week 62
  Changes from baseline in POEM
EuroQol Five Dimensions Questionnaire (EQ-5D) | up to week 62
  Changes from baseline in EQ-5D
Pharmacokinetics parameters | up to week 62
  Trough concentration and exposure of CM310
Immunogenicity | up to week 62
  Detection of anti-drug antibody (ADA) and neutralizing antibody (Nab)

CONTACTS AND LOCATIONS:
Overall Officials: jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's hospital, Beijing, China